CLINICAL TRIAL: NCT00710359
Title: Cobalamin Status in Young Children With Gastrointestinal Symptoms or Feeding Problems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Collaborators: Norwegian Foundation for Health and Rehabilitation (Other); Foundation to Promote Research into Functional Vitamin B12 Deficiency, Bergen, Norway (Other)
Responsible Party: Anne-Lise Bjørke Monsen, Haukeland University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 19157
Record Dates: First submitted 2008-07-02; First posted 2008-07-04 (Estimated); Last update posted 2010-08-16 (Estimated); Status verified 2010-08

CONDITIONS: Vitamin B 12 Deficiency
Keywords: Cobalamin deficiency; Infant; Nutrition; Cobalamin supplementation; Feeding problems; Gastrointestinal symptoms
MeSH Terms: conditions — Vitamin B 12 Deficiency | interventions — Hydroxocobalamin; Vitamin B 12; Vitamin B Complex

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): 400 µg hydroxycobalamin (Vitamin B12 Depot, Nycomed Pharma) given as a single intramuscular injection. The syringe is covered so it is impossible to see whether or not it contains any substance.
  Interventions: Dietary Supplement: Hydroxycobalamin (Vitamin B12 Depot, Nycomed Pharma)
- 2 (Sham Comparator): The controls receive an intramuscular "injection", however, it is only an introduction of the needle into the muscle, but no injections are given. The syringe is covered so it is impossible to see whether or not it contains any substance.
  Interventions: Dietary Supplement: Hydroxycobalamin (Vitamin B12 Depot, Nycomed Pharma)

INTERVENTIONS:
Dietary Supplement: Hydroxycobalamin (Vitamin B12 Depot, Nycomed Pharma) — 400 µg hydroxycobalamin (Vitamin B12 Depot, Nycomed Pharma), as a single intramuscular injection
  Other Names: Vitamin B12; Cobalamin; B vitamins

SUMMARY:
During fetal life and infancy, an adequate cobalamin status is important for normal growth and central nervous system development. During the last years we have detected cobalamin deficiency in a number of infants admitted to the Pediatric Department with various symptoms, including neurological symptoms and feeding problems. Cobalamin treatment is given to the infants with biochemical cobalamin deficiency, and leads to loss of symptoms and in improved physical condition.

In this study we want to establish the prevalence of cobalamin deficiency in infants with gastrointestinal symptoms and/or feeding problems. Cobalamin status will be investigated in all children aged 8 months and younger, admitted to the Pediatric Department with these symptoms. In a randomised intervention trial we will evaluate the effect of cobalamin supplementation in children with these symptoms and metabolic evidence of impaired cobalamin status.

Study hypothesis: Cobalamin treatment given to the infants with biochemical cobalamin deficiency, will lead to loss of symptoms and in improved physical condition.

ELIGIBILITY:
Inclusion Criteria:

* Children below 8 months of age
* Clinical diagnosis or symptoms: feeding problems and/or gastrointestinal symptoms

Exclusion Criteria:

* Children with syndromic disease

Max Age: 8 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2008-04; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Outcome Measure: Changes in cobalamin and folate status, including metabolic markers, hematological parameters, growth parameters, symptom and neurological evaluation | Reevalutation after 4 weeks

SECONDARY OUTCOMES:
Maternal evaluation of changes in infant behaviour and symptoms | After 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Lise Bjørke Monsen, M.D., Ph.D., Principal Investigator — Laboratory of Clinical Biochemistry, Haukeland University Hospital, N-5021 Bergen, Norway; Per Magne Ueland, M.D., Ph.D., Study Director — Department of Internal Medicine, University of Bergen, 5021 Armauer Hanssen Hus, Bergen, NORWAY
Locations (1):
- Department of Pediatrics, Haukeland University Hospital, Bergen, Norway

REFERENCES:
- [Background] Rosenblatt DS, Whitehead VM. Cobalamin and folate deficiency: acquired and hereditary disorders in children. Semin Hematol. 1999 Jan;36(1):19-34. PMID 9930566
- [Background] Bjorke Monsen AL, Ueland PM, Vollset SE, Guttormsen AB, Markestad T, Solheim E, Refsum H. Determinants of cobalamin status in newborns. Pediatrics. 2001 Sep;108(3):624-30. doi: 10.1542/peds.108.3.624. PMID 11533328
- [Background] Wulffraat NM, De Schryver J, Bruin M, Pinxteren-Nagler E, van Dijken PJ. Failure to thrive is an early symptom of the imerslund Grasbeck syndrome. Am J Pediatr Hematol Oncol. 1994 May;16(2):177-80. PMID 8166372
- [Background] Monsen AL, Refsum H, Markestad T, Ueland PM. Cobalamin status and its biochemical markers methylmalonic acid and homocysteine in different age groups from 4 days to 19 years. Clin Chem. 2003 Dec;49(12):2067-75. doi: 10.1373/clinchem.2003.019869. PMID 14633879
- [Background] Bjorke-Monsen AL, Torsvik I, Saetran H, Markestad T, Ueland PM. Common metabolic profile in infants indicating impaired cobalamin status responds to cobalamin supplementation. Pediatrics. 2008 Jul;122(1):83-91. doi: 10.1542/peds.2007-2716. PMID 18595990
- [Derived] Torsvik I, Ueland PM, Markestad T, Bjorke-Monsen AL. Cobalamin supplementation improves motor development and regurgitations in infants: results from a randomized intervention study. Am J Clin Nutr. 2013 Nov;98(5):1233-40. doi: 10.3945/ajcn.113.061549. Epub 2013 Sep 11. PMID 24025626